CLINICAL TRIAL: NCT04012710
Title: Transvaginal Natural Orifice Transluminal Endoscopic Surgery- A New Approach to Salpingo-oophorectomy
Brief Title: vNOTES for Salpingo-oophorectomy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Collaborators: Assuta Medical Center (Other)
Responsible Party: Principal Investigator, Dr. Aya Mohr-Sasson, Principle Investigator, Sheba Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 32-19-ASMC
Record Dates: First submitted 2019-07-07; First posted 2019-07-09 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Surgery
Keywords: Transvaginal natural orifice transluminal endoscopic surgery; Salpingo-oophorectomy; Laparoscopy
MeSH Terms: interventions — Laparoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Laparoscopy (Active Comparator): Abdominal conventional laparoscopy for salpingo-oophorectomy
  Interventions: Procedure: Laparoscopy
- vNOTES (Active Comparator): Transvaginal natural orifice transluminal endoscopic surgery for salpingo-oophorectomy
  Interventions: Procedure: vNOTES

INTERVENTIONS:
Procedure: Laparoscopy — Conventional abdominal laparoscopy
  Arms: Laparoscopy
Procedure: vNOTES — Transvaginal natural orifice transluminal endoscopic surgery for salpingo-oophorectomy
  Arms: vNOTES

SUMMARY:
The aim of this study is to compare the common approach of laparoscopy for bilateral salpingo - oophorectomy to a new approach via transvaginal natural orifice transluminal endoscopic surgery (vNOTES).

DETAILED DESCRIPTION:
Natural Orifice Transluminal Endoscopic Surgery (NOTES) is an emerging field in minimally invasive surgery. NOTES can be performed via a variety of approaches, including through the stomach, esophagus, bladder, and rectum, but the majority of cases have been performed transvaginally (vNOTES).

The vNOTES technique includes conventional, laparoscopic instruments that are inserted through a single-port device that enables the insertion of 1 10-mm trocar, and 4 5-mm trocars. The operation in carried out placing the patient in the lithotomy position. After completing general anaesthesia, a 2.5-cm posterior colpotomy is made. The pouch of Douglas is opened and the transvaginal natural orifice transluminal endoscopic surgery (vNOTES) port is inserted transvaginally. A pneumoperitoneum is created, and the pelvic cavity, including the uterus and the adnexa is demonstrated. Only then, the conventional laparoscopic instruments are inserted.

By incorporating the advantages of endoscopic surgery, the vNOTES approach avoids abdominal wall wounds and trocar-related complications, including reducing post operation pain. Moreover, recent studies report, shorter hospital stay, improved visibility, and the possibility to circumvent extensive lysis of adhesion to reach the pelvic cavity. It should be mentioned that operative risks such as : anesthesia complications, excessive blood loss, damage to near organs ( intestines or bladder), and vasculature damage exists in both conventional laparoscopy and vNOTES approach.

vNOTES technique has been used for hysterectomy and was proven to be just as good as laparoscopy with the advantage of daycare surgery. The use of vNOTES for salpingo-oophorectomy without concomitant hysterectomy has been questioned due to challenging accessibility. To the best of our knowledge, data concerning the experience using this technique for salpingo-oophorectomy is scarce and based on few published case-reports.

Therefore, the aim of this study is to compare the common approach of laparoscopy for bilateral salpingo - oophorectomy to a new approach via transvaginal natural orifice transluminal endoscopic surgery (vNOTES).

Material and methods

This is a randomized prospective study including women admitted electively to a single care center for bilateral salpingo-oophorectomy due to benign indication. Women that will be found to fit inclusion criteria will get by the research team explanation on both techniques. After giving informed consent, all women will be allocated to one of two operative techniques by en-block randomization:

1. Laparoscopy
2. vNOTES

Both operations will be done by a single highly skilled operator. All women will sign informed consent before admitted to operation room. Patient's demographics, characteristics, perioperative, operative and post-operative data will be collected from medical records. Data will be coded in order to save confidentiality ( each serial number will identify a patient. The list of serial numbers that fits each identification number will be available only for the principle investigator ).

ELIGIBILITY:
Inclusion Criteria:

* Elective surgery
* Benign indication for surgery

Exclusion Criteria:

* Severe endometriosis
* Past pelvic operations
* Suspected malignancy
* Combined planned hysterectomy
* Recurrent Pelvic Inflammatory disease (PID)
* Vaginal anomaly

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Only women planned to undergo bilateral salpingo-oophorectomy
  .
Enrollment: 100 (Estimated)
Dates: Start 2025-07-03 (Estimated); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Intra - Operative complication rate | Intra - Operative
  Complications during operation as a compound outcome including - bleeding. damage to neer organs and vasculature damage

SECONDARY OUTCOMES:
Woman satisfaction rate post operation | Estimated on post operation day -1- through study completion, an average of 1 year
  Satisfaction rate estimated by VAS -Visual Analogue Scale - A numeric satisfactory rating scale scoring 0 to 10, while 0 is not satisfied at all and 10 is highly satisfied .

CONTACTS AND LOCATIONS:
Overall Officials: Aya Mohr-Sasson, Principal Investigator — Assuta Medical Center, Israel
Locations (1):
- Aya Mohr Sasson, Ramat Gan, Please Select, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Jallad K, Walters MD. Natural Orifice Transluminal Endoscopic Surgery (NOTES) in Gynecology. Clin Obstet Gynecol. 2017 Jun;60(2):324-329. doi: 10.1097/GRF.0000000000000280. PMID 28221179
- [Result] Tantitamit T, Lee CL. Application of Sentinel Lymph Node Technique to Transvaginal Natural Orifices Transluminal Endoscopic Surgery in Endometrial Cancer. J Minim Invasive Gynecol. 2019 Jul-Aug;26(5):949-953. doi: 10.1016/j.jmig.2018.10.001. Epub 2018 Oct 5. PMID 30296476
- [Result] Boesen L, Meisner S, Vilmann P, Jorgensen LN, Rosenberg J, Donatsky AM. [Transvaginal hybrid natural orifice transluminal endoscopic surgery cholecystectomy]. Ugeskr Laeger. 2016 Jan 25;178(4):V06150482. Danish. PMID 26815719
- [Result] Hiep PN, Thien HH, Vu PA, Thanh PH, Xuan NT. Natural orifice transluminal endoscopic surgery for colorectal cancer. BJS Open. 2017 May 24;1(1):24-29. doi: 10.1002/bjs5.4. eCollection 2017 Feb. PMID 29951602
- [Result] Baekelandt J. Transvaginal natural orifice transluminal endoscopic surgery: a new approach to ovarian cystectomy. Fertil Steril. 2018 Feb;109(2):366. doi: 10.1016/j.fertnstert.2017.10.037. Epub 2017 Dec 13. PMID 29246560
- [Result] Baekelandt J, De Mulder PA, Le Roy I, Mathieu C, Laenen A, Enzlin P, Weyers S, Mol BW, Bosteels JJ. Postoperative outcomes and quality of life following hysterectomy by natural orifice transluminal endoscopic surgery (NOTES) compared to laparoscopy in women with a non-prolapsed uterus and benign gynaecological disease: a systematic review and meta-analysis. Eur J Obstet Gynecol Reprod Biol. 2017 Jan;208:6-15. doi: 10.1016/j.ejogrb.2016.10.044. Epub 2016 Oct 29. PMID 27880893
- [Result] Baekelandt JF, De Mulder PA, Le Roy I, Mathieu C, Laenen A, Enzlin P, Weyers S, Mol B, Bosteels J. Hysterectomy by transvaginal natural orifice transluminal endoscopic surgery versus laparoscopy as a day-care procedure: a randomised controlled trial. BJOG. 2019 Jan;126(1):105-113. doi: 10.1111/1471-0528.15504. PMID 30325565
- [Result] Baekelandt JF, De Mulder PA, Le Roy I, Mathieu C, Laenen A, Enzlin P, Weyers S, Mol BWJ, Bosteels JJA. Transvaginal natural orifice transluminal endoscopic surgery (vNOTES) adnexectomy for benign pathology compared with laparoscopic excision (NOTABLE): a protocol for a randomised controlled trial. BMJ Open. 2018 Jan 10;8(1):e018059. doi: 10.1136/bmjopen-2017-018059. PMID 29326183
- [Result] Terzi H, Turkay U, Uzun ND, Salici M. Hysterectomy and salpingo-oophorectomy by transvaginal natural orifice transluminal endoscopic surgery (V-NOTES) assisted by an umbilical camera: Case report and new hybrid technique in gynecology. Int J Surg Case Rep. 2018;51:349-351. doi: 10.1016/j.ijscr.2018.08.053. Epub 2018 Sep 5. PMID 30248628